CLINICAL TRIAL: NCT05304533
Title: An Open-label, 3-Arm, Parallel Design Pharmacokinetic Interaction Study Between MYK-224 and Cytochrome P450 3A4 Inhibitors Itraconazole and Verapamil in Healthy Participants
Brief Title: A Study to Assess the Drug Interaction Between MYK-224 and Itraconazole and Verapamil in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CV029-005
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Healthy Participants
Keywords: MYK-224; Itraconazole; Verapamil
MeSH Terms: interventions — Itraconazole; Verapamil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: MYK-224 (Experimental)
  Interventions: Drug: MYK-224
- Arm 2: MYK-224 + Itraconazole (Experimental)
  Interventions: Drug: MYK-224; Drug: Itraconazole
- Arm 3: MYK-224 + Verapamil (Experimental)
  Interventions: Drug: MYK-224; Drug: Verapamil

INTERVENTIONS:
Drug: MYK-224 — Specified dose on specified days
  Other Names: BMS-986435
Drug: Itraconazole — Specified dose on specified days
  Arms: Arm 2: MYK-224 + Itraconazole
Drug: Verapamil — Specified dose on specified days
  Arms: Arm 3: MYK-224 + Verapamil

SUMMARY:
The purpose of this study is to evaluate the effect of co-administration of itraconazole or verapamil on the drug levels of MYK-224 in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18 and 30 kg/m^2, inclusive
* Healthy as determined by medical history, physical examination, vital signs, 12-lead electrocardiogram and routine laboratory assessments
* Adequate acoustic windows to enable accurate transthoracic echocardiographic assessment
* Left Ventricular Ejection Fraction (LVEF) ≥60% at screening and ≥55% prior to MYK-224 dosing

Exclusion Criteria:

* Any acute or chronic medical illness
* History of dizziness and/or recurrent headaches
* History of heart disease

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to 36 days
Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration (AUC[0-T]) | Up to 36 days
Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC[INF]) | Up to 36 days

SECONDARY OUTCOMES:
Time of maximum observed plasma concentration (Tmax) | Up to 36 days
Apparent terminal plasma half-life (T-HALF) | Up to 36 days
Apparent total body clearance (CLT/F) | Up to 36 days
Number of participants with adverse events (AEs) | Up to 52 days
Number of participants with serious adverse events (SAEs) | Up to 52 days
Number of participants with adverse events leading to discontinuation | Up to 52 days
Number of participants with vital sign abnormalities | Up to 52 days
Number of participants with electrocardiogram (ECG) abnormalities | Up to 52 days
Measurement of left ventricular ejection fraction (LVEF) | Up to 52 days
Measurement of left ventricular outflow tract velocity time integral (LVOT-VTI) | Up to 52 days
Measurement of left ventricular fractional shortening (LVFS) | Up to 52 days
Measurement of left ventricular global longitudinal strain (LV GLS) | Up to 52 days
Measurement of left ventricle stroke volume (LVSV) | Up to 52 days
Number of participants with physical exam abnormalities | Up to 52 days
Number of participants with clinical laboratory abnormalities | Up to 52 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Dallas, Texas, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/us/en/home.html